CLINICAL TRIAL: NCT01661465
Title: Routine Clinical Screening for Substance Use Disorders in the Emergency Room Setting
Status: Terminated | Type: Observational
Why Stopped: The Principal Investigator left the site.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Cheryl McCullumsmith, Division Director, Hospital Psychiatry, University of Alabama at Birmingham
Other Study IDs: X110422001
Record Dates: First submitted 2012-08-07; First posted 2012-08-09 (Estimated); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To ensure consistent documentation of alcohol and substance use, the emergency medicine is initiating a new standard of care for substance use screening: the use of a brief self-evaluation questionnaire on alcohol, tobacco and illicit substance use to be completed in triage. This questionnaire will allow emergency medicine patients presenting to the emergency room. This study will also review medical records after one year of the index emergency room visit to establish rates or re-presentation and hospitalization correlated with different substance use.

DETAILED DESCRIPTION:
Screening for alcohol use and substances of abuse in the emergency and trauma settings is critical for both effective current treatment of the presenting clinical issue and prevention of future incidents. Identification, engagement and treatment of substance use disorders decreased trauma and emergency department visits and medical comorbidities (Bertholet et al., 2005; Kaner et al., 2007). To ensure consistent documentation of alcohol and substance use, the emergency medicine is initiating a new standard of care for substance use screening: the use of a brief self-evaluation questionnaire on alcohol, tobacco and illicit substance use to be completed in triage. This questionnaire will allow emergency medicine patients presenting to the emergency room. This research study will perform a chart review on all self-evaluation questionnaires on alcohol, tobacco and substance use to determine the prevalence of use of specific substances in this patient population and associated demographic predictors and medical comorbidities. This study will also review medical records after one year of the index emergency room visit to establish rates or re-presentation and hospitalization correlated with different substance use.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete a questionnaire

Exclusion Criteria:

* Younger than 19 Unable or unwilling to complete a self-assessment form written in English Prisoners

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting to University Hospital Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 9212 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with re-presentation of drug or alcohol abuse 1 year after initial presentation to Emergency Department | baseline to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama Birmingham, Birmingham, Alabama, United States